CLINICAL TRIAL: NCT06936033
Title: The Effects of Kinesiology Taping on Joint Stability During Descending Stairs in Patients With Acute Ankle Injuries
Brief Title: Kinesiology Taping and Ankle Stability in Acute Injuries During Stair Descent
Acronym: KTAS-SD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo University (Other)
Responsible Party: Principal Investigator, ye wei, Principal Investigator, Ningbo University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: TY2025004
Record Dates: First submitted 2025-03-05; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-09

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KT Group: Kinesio Taping for Acute Ankle Injuries (Experimental): This arm involves the application of Kinesio Taping (KT) to participants with acute ankle injuries. The KT intervention uses Kinesio®Tex GOLD™ tape, applied with specific tension and directional control to stabilize the ankle joint, limit excessive inversion/eversion, and enhance proprioception.
  This study used a control experiment between the ST group without Kinesio Taping intervention and the KT group with Kinesio Taping intervention. The stability, gait analysis, and impact force of the ankle lower limb movement in patients with acute ankle injury were compared before and after Kinesio Taping and without Kinesio Taping.
  Interventions: Other: Kinesiology taping
- ST Group: no Kinesio Taping (No Intervention)

INTERVENTIONS:
Other: Kinesiology taping — This study used Kinesio taping as an intervention to compare the biomechanical effects of stair descent in patients with acute ankle injuries before and after taping. Participants participated in two intervention conditions: the KT experimental group (Kinetoscopy taping) and the ST control group (no Kinesio taping), and each condition performed 20 separate stair descent tests.
  Arms: KT Group: Kinesio Taping for Acute Ankle Injuries

SUMMARY:
Background: Acute ankle injuries are common in sports and daily activities. Kinesiology taping enhances lower limb motion patterns, joint stability, and balance during descending stair activity in such patients. The objective of this study was to conduct a comparative analysis of the biomechanical impacts exerted by a KT group and an ST group on the lower limbs of patients with acute ankle injuries while descending stairs.

Methods: The study included 27 participants with acute ankle injuries, who underwent biomechanical assessment under both KT and ST conditions. An integrated Vicon motion capture system, AMTI force platform, and electromyography (EMG) sensors were utilized to comprehensively evaluate biomechanical performance. Participants completed 20 descending stair trials under each condition, with joint stiffness, center of mass (COM), and bone displacement identified as key metrics for assessing stability. Statistical analyses, including paired t-tests and statistical parametric mapping (SPM1D), were employed to identify significant biomechanical differences between the two conditions.

DETAILED DESCRIPTION:
Background Acute ankle injuries (ATIs) are among the most common injuries experienced by athletes, particularly in sports like football, basketball, and running. Research indicates that acute ankle injuries, particularly those sustained during high-intensity sports, are associated with an increased risk of long-term functional instability in athletes. Maresh reviewed the functional instability that may result after ankle ligament injury and emphasized the importance of early intervention and effective rehabilitation of acute ankle injuries. Biomechanical studies have further revealed the impact of acute ankle injuries on the kinetics stability of the lower limbs. Acute ankle injuries may affect the motion patterns of the ankle joint and its adjacent joints (knee, hip), resulting in decreased stability during motion and increased risk of other injuries. In addition, Wang, et al. studied the biomechanics of the knee joint through step width and proposed the idea of joints working together during motion, which is also of great significance for the understanding of acute ankle joint injuries. To minimize the risk of acute ankle injuries, Willson conducted a systematic review highlighting several prevention strategies. These include the use of ankle braces by athletes, careful selection of appropriate sports footwear, and the optimization of training programs. Together, these measures aim to effectively prevent and reduce the incidence of such injuries. Therefore, it is important to explore theoretical and practical significance to explore how to improve the stability of the ankle joint through effective means, reduce the risk of sports injuries, and improve body stability.

Among the many experimental research publications that explore the kinematic characteristics, kinetics mechanisms, and joint stiffness changes in patients with acute ankle injuries during climbing and descending stairs, multiple studies have explored the impact of different factors on ankle joint stability. Research has revealed that there is a close relationship between changes in ankle flexion and extension angles and gait efficiency and stability. Wang et al. focused their research perspective on the impact of step width on the biomechanical properties of the knee joint and emphasized that the synergy between the ankle joint and the knee joint plays an indispensable role in maintaining overall stability. Protopapadaki et al. conducted a comprehensive analysis of the changes in flexion-extension angles and moments of the ankle joint during ascending and descending stair walking. They highlighted that a greater ankle flexion angle during descending stair actions may significantly elevate the risk of ankle joint injury. The study by Riener et al. focused on the maximum flexion angle of the knee joint when descending stairs and found that there is a significant correlation between the angle change of the knee joint, the range of motion, and the load borne by the ankle joint. Novak and Brouwer analyzed the fluctuations of joint moments during the process of ascending and descending stairs, revealing that the increase in ankle joint load in the elderly may induce the risk of injury. The study by Gill et al. further explored the intrinsic connection between trunk tension and postural balance, emphasizing the important role of coordination between the trunk and lower limbs in maintaining ankle joint stability. Major et al. examined the impact of prosthetic foot stiffness on gait and muscle function and pointed out that similar stiffness changes may also have a profound impact on the ankle joint stability of healthy individuals.

Kinesiology Taping (K-Taping), as a technology commonly used in sports medicine and rehabilitation treatment and has been widely used around the world in recent years. Through its unique elastic material design and fitting technique, k-taping provides additional support and protection for muscles and joints without restricting joint motion, thereby enhancing muscle contraction, improving endurance, reducing tremors and pain, and ultimately improving joint stability. However, although k-taping is increasingly used in the field of sports medicine, its specific impact on the stability and motion efficiency of specific joints (such as ankle joints) still requires further in-depth analysis. Research by Biz et al. revealed the positive impact of k-taping on the range of motion of the ankle joints during running activities, helping to improve joint stability and overall sports performance. The study by Wikstrom et al. emphasized the significant role of k-taping in adjusting muscle activation patterns and joint moments in patients with acute ankle injuries, especially in controlling ankle eversion moments. In the context of ascending and descending stairs, research by Paquette's team demonstrates that k-taping can reduce the load on the ankle joint, optimizing the joint motion trajectory, and consequently lower the risk of injury. Aytar et al. further explored the effect of k-taping on muscle force and joint stiffness and found that it can significantly improve muscle force in the injured area and increase joint stiffness, thereby enhancing the patient's motion ability and stability. Research by Ellis 's team revealed the unique role of k-taping in coordinating the kinematic patterns of the ankle joint and knee joint, helping to reduce the burden on the ankle joint and improve overall motion coordination. Halseth et al. further verified the positive effect of k-taping in expanding the range of ankle joint motion and improving muscle activation levels, providing strong support for patient rehabilitation. At the same time, research by Lee 's team observed that k-taping has a significant effect in improving ankle joint stability and muscle activation levels, especially in kinetics motions. In addition, the research by Fayson et al. also showed that k-taping can improve the joint stiffness and muscle force output of the ankle joint, providing an effective means for patients with acute ankle injuries to improve lower limb stability and reduce the risk of reinjury.

The aim of this study was to explore the effects of KT and ST on the biomechanics of patients with acute injuries using a descending stairs task. The investingactors hypothesized that through the intervention of intramuscular patching, the stability of the ankle joint of k-taping patients would be strengthened, which would help to enhance the stability of the ankle joint and thereby better maintain balance during the process of walking down descending stairs.

Methods The study used a randomized crossover design to investigate the biomechanical effects of muscle efficiency patches while walking down descending stairs. Twenty-seven subjects with acute ankle injuries participated in the study. Subjects participated in two sets of intervention conditions: the KT experimental group (exercise Kinesio tape) and the ST control group (no Kinesio tape), with three separate descending stairs tests for each condition. The biomechanical performance of the acutely injured subjects during a descending stairs task was compared with the ST group focusing on lower extremity motion stability and gait analysis, impact forces, etc. A Vicon Motion Capture System, featuring eight cameras, was integrated with the AMTI Force Platform to concurrently gather biomechanical data. This data encompassed joint angles, moments, and power during the pre-weight-bearing, mid-stance, and push-off phases of the affected limb, as documented in reference. Additionally, Electromyography (EMG) equipment from Delays, Boston, MA, USA, was employed to assess muscle activation patterns, as described in reference.

Participants In this study, a priori efficacy analyses were conducted using G*Power (version: 3.1.9.7; Henry Düsseldorf University, Düsseldorf, Germany) software to determine the sample size required for the experimental design. The findings demonstrated that a minimum sample size of 27 participants was necessary to attain a moderate effect size of 0.50. By completing the AOFAS (American Orthopaedical Foot & Ankle Society) Ankle-Hindfoot Scale as well as the VAS scale, 27 subjects with acute ankle injuries from Ningbo University were selected (Age: 18.30±25.80 years; Height: 162.45±185.14 cm; Weight: 60.20±85.05 kg). Participants were chosen according to the following criteria: Subjects had experienced at least one acute sprain of the ankle joint. Those who experienced symptoms of pain and instability during daily activities or sports. No other serious diseases affect the function of the lower limbs (e.g., arthritis, severe knee lesions, etc.). AOFAS < 80 points and VAS ≤ 3 on the affected side. The onset of injury is usually limited to 7 days to ensure that it is in the acute phase. Participants maintained a steady level of daily activity during the study period. Exclusion Criteria: History of severe structural injury or surgery to the ankle (e.g., ligament reconstruction surgery, arthroscopic surgery, etc.). Presence of neuromuscular disease, or women during pregnancy. Allergy to muscle patch materials or history of skin disease. Ankle-related surgery or rehabilitation within the last 6 months. Before the initiation of data collection, all participants provided their written informed consent. Additionally, the study received ethical approval from the Ethics Committee of Ningbo University, ensuring that the research adhered to the highest ethical standards (Approval Number: TY2025004).

Data collection procedures All the experimental tests were conducted within the Exercise Biomechanics Laboratory of the Institute of Greater Health, situated at Ningbo University in Ningbo, China. The laboratory is outfitted with a sophisticated Vicon motion capture system (Oxford Metrics Ltd, Oxford, UK). This state-of-the-art system incorporates eight high-precision cameras, which were employed to accurately record three-dimensional motion data as the participants were engaged in the activity of descending stairs. The sampling frequency for the Vicon motion capture system (Oxford Metrics Ltd, Oxford, UK) was configured at 200 Hz, and the system underwent meticulous calibration before each test to ensure precise measurements of joint kinematics and motion. Calibration included positioning reflective markers at predefined locations within the capture area and adjusting the cameras for optimal alignment and accuracy. This procedure was repeated at the start of each data collection session to maintain consistency in measurements. The force platform, sourced from AMTI in Watertown, Massachusetts, USA, was configured with a sampling frequency of 1000 Hz. This specific frequency setting was deliberately chosen to ensure a precise and detailed recording of ground reaction forces as the participants descended the stairs. Through this high sampling rate, any subtle variations and dynamic changes in the forces exerted on the ground during the stair - descent process could be accurately captured and analyzed. The two systems were precisely synchronized to ensure seamless data collection. The initial contact point during the stair descent was determined based on a specific criterion. It was identified when the vertical ground reaction force registered a value exceeding 10 Nm. This standardized method of identifying the initial contact point allowed for consistent and accurate data analysis, facilitating a more in-depth understanding of the biomechanical processes involved in stair descent. The AMTI force platform was also calibrated before each test following the manufacturer's instructions, which involved applying a known load to verify and adjust the force output for accurate readings.

All participants wore standardized tight-fitting clothing and remained barefoot to ensure the visibility of body markers used for motion capture. Anthropometric measurements, including height, weight, and leg length, were documented. A total of 38 markers, each 14 mm in diameter, were placed on the lower limbs and torso following the Opensim Gait-2392 model. Reflective markers were placed on specific anatomical landmarks, The placement of EMG sensors adhered to the SENIAM guidelines, with eight sensors positioned on the muscle groups of the soleus, medial and lateral gastrocnemius, tibialis anterior, rectus femoris, and medial and lateral vastus muscles, The EMG system, used to capture muscle activation data, underwent calibration using standardized protocols, which included verifying sensor signal accuracy and optimizing the system to minimize noise and ensure consistent data acquisition. To enhance signal quality, skin preparation techniques such as shaving and the application of cleansing gels were performed. The EMG system's reliability in recording muscle activity during exercise has been validated in previous studies.

The Vicon motion capture system, the AMTI force platform, and the EMG system were synchronized to enable integrated data acquisition. Before starting the experiment, a static calibration procedure was conducted to support the subsequent creation of manikins. Participants were first introduced to the experimental conditions and procedures. During static data collection, participants stood on the force platform with their feet aligned parallel to the y-axis, arms extended at a 45° angle from their sides, and gaze fixed forward. This posture was maintained until the static data collection was complete. The RLA gait analysis method of Rancho Los Amigos (RLA) Medical Center, California, USA was used.

In this study, 5 cm wide KinesioTaping (Kinesio®Tex GOLDTM) were applied to the participants, which were characterized as being able to be stretched to 140% of their original length. The K-Taping technique was applied following the methodology outlined by Jackson et al. This experiment used a randomized grouping and crossover design to divide the subjects into KT group and ST group. KT group used K-Taping (four tapes were applied to the foot (the foot was kept in dorsiflexion at 90 degrees) to provide support and stability. The first tape was anchored at the midpoint below the heel bone, with 20% tension applied at both ends to extend up the sides of the heel and talus, and slightly rotate over the tibialis anterior muscle to minimize side-to-side ankle rotation; the second tape was applied laterally at 50% tension to the lateral heel bone, extending around the heel to the medial first metatarsal bone to limit foot rotation; and the third tape, again at 50% tension, was applied to the medial talus, wrapped around the heel, and wrapped around the medial first metatarsal bone to limit foot rotation.

The third tape, also at 50% tension, starts at the medial talus, wraps around the heel and over the fourth and fifth metatarsals to further enhance plantar stability; the fourth tape is anchored from the navicular bone, wraps around the plantar foot to the lateral cuneiform bone at 20% tension, then increases to 80% tension around the Achilles tendon posteriorly to anchor it to the lateral ankle, and finally extends at 50% tension to cover the first and second metatarsal bones and wraps around the entire area. (This method of applying the patch is suitable for the protection and support needs in sports through the precise distribution of tension and directional control to fully limit the rotation and turning of the foot, and at the same time to strengthen the stability of the ankle joint and the sole of the foot) In ST group, the muscle patch was not used, and only the routine test was performed. The experimental task was a descending stairs test, which was done on a four-step staircase (each step was 300 mm in length, 900 mm in width, and 170 mm in height), and subjects were asked to complete the task of descending the staircase 20 times with a natural gait in each experimental condition. All subjects were required to be barefoot. The test was divided into two conditions, KT group and ST group, with a 5 to 10-minute break between conditions to avoid fatigue interference. Kinematic data, descending stairs time and gait stability were recorded during the experiment, and subjective perception was collected. At the end of the experiment, the muscle patch was removed, the patch site was cleaned, and the data were organized and backed up to provide a basis for subsequent analysis. The safety of the subjects was ensured throughout the experiment to avoid accidents.

To gather biomechanical data and ensure that subjects accurately complete the descending stairs task, the study will first schedule subjects to perform a standardized warm-up to ensure that the lower extremity muscles are fully activated. Prior to the start of the test, subjects familiarized themselves with the descending stairs maneuver by practicing and marking clear start and end positions on the stairs to ensure a consistent pace for each test. Data for each test was collected using a high-precision motion capture system and force platform, mainly involving changes in knee and ankle joint angles, EMG signals and joint forces. If the subject failed to complete the motion or the motion was not standardized, it was considered a failure and was not counted in the data analysis.

High-speed biplane fluorescence fluoroscopy imaging system High-speed biplane fluorescence fluoroscopy imaging system (DFIS) comprises a motion fluoroscopy system and a data resolution system. The former consists of two high-voltage emitters and light sources, two movable robotic arms with fluorescence receivers and intensifiers, and two high-speed cameras. The distances between the 2 high-voltage emitters and receivers are 132.2 cm and 128.6 cm, respectively, with an angle of 119.6° between the image receivers; the shooting parameters were set as follows: a voltage of 60 KV, a current of 63 MA, a shooting frequency of 100 Hz, an exposure speed of 1/1000 s, and an image resolution of 1024 * 1024 pixels.

The environment calibration file generated by XMAlab was imported into Rhinoceros software for further processing. Its modeling module was used to reconstruct the shooting space and restore the relative positions of the two pairs of fluorescence emitters and image receivers in the virtual space; meanwhile, the aberration-calibrated foot and ankle X-ray images and the 3D models of the tibia, the talus, and the calcaneus were imported. The coordinate systems of the tibia, talus and heel were established according to previous standards, and the tibial-posterior, lateral-medial and superior-inferior directions corresponded to the x-axis, y-axis and z-axis, respectively, whereas plantar/dorsiflexion, inversion/eversion, and internal/external rotation were defined as the motion around the tibial-posterior, lateral-medial and superior-inferior axes, respectively. The imported skeletal models were then rotated and translated in the 3D space reconstructed by the Rhinoceros software until the skeletal projections in each frame matched the skeletal contours in the fluoroscopic images.

The 6DOF data of the superior talar joint (talus versus tibia) and the inferior talar joint (heel versus talus) were calculated using the Coordinate System Calculation Plug-in Rhinoceros, which includes kinematic data in three translational (tibial-posterior, lateral-medial and superior-inferior) and three rotational (plantar/dorsiflexion, inversion/eversion, and internal/external rotation) directions. Positive values represent outward, forward, and upward translation of the talus relative to the tibia (heel relative to the talus), as well as dorsiflexion, inversion, and internal rotation; negative values represent inward, backward, and downward translation, as well as plantarflexion, eversion, and external rotation.

Kinematic and kinetics data collected from Vicon were exported to C3D file format, then converted to a coordinate system, low pass filtered, data extracted and formatted for kinematic and ground reaction force (GRF) data using MATLAB (MathWorks, Massachusetts, USA). The C3D files were converted to TRC and MOT file formats using MATLAB and subsequently imported into OpenSim (Stanford University, Stanford, CA, USA) to compute biomechanical parameters. Musculoskeletal simulations were conducted using a model with 23 degrees of freedom and 92 muscle actuators. OpenSim's scaling tools enabled the creation of subject-specific musculoskeletal models by adapting a generic model to align with individual body dimensions. These scaling adjustments were applied to segment lengths, segment inertia properties, and muscle attachment points. Muscle origin and insertion points, along with muscle moment arms, were tailored to match each participant's limb dimensions. Residual moments in the frontal and lateral planes were minimized during the simulation process. The inverse kinematics tool used a weighted least squares optimization to calculate joint angles, reducing discrepancies between model-generated and experimental marker positions. The inverse kinetics tool computed joint moments for each degree of freedom, and joint power was determined by multiplying the angular velocity by the joint moment at each time step.

A static optimization algorithm was used to estimate muscle activation and muscle force, and the results were compared to surface EMG activity recorded during experiments to validate the model. The signal-to-noise ratio was optimized by performing residual analysis on a subset of data from previous studies. Kinematic and kinetic data were filtered using a fourth-order zero-lag Butterworth low-pass filter with cutoff frequencies of 12 and 20 Hz, respectively. Surface EMG signals were preprocessed by band-pass filtering with a fourth-order Butterworth filter in the frequency range of 10-400 Hz. This was followed by full-wave rectification and low-pass filtering with a cutoff frequency of 6 Hz. Additionally, the EMG signals were normalized by dividing the EMG amplitude by the maximum root-mean-square (RMS) amplitude. The signals were further normalized using the maximum voluntary contraction (MVC) to determine the activation level of each muscle. The muscle activation results recorded by the EMG sensors were compared with those simulated by the musculoskeletal model to evaluate the model's validity and accuracy.

Model accuracy was enhanced using specific equations and plug-ins in OpenSim. Joint angles were calculated using an inverse kinematics algorithm, while joint moments were determined using an inverse kinetic algorithm. A residual reduction algorithm was also applied to address kinetic inconsistencies in the model. The inverse kinematics tool optimized joint angle computations by employing a weighted least squares approach to minimize discrepancies between model-predicted and experimental marker positions. Joint moments were computed for each degree of freedom in the model, and joint power was subsequently calculated as the product of angular velocity and joint moment at each time point.

Statistical Analysis Data from the lower staircase trials were analyzed using a paired samples t-test (with a significance level of 0.05 and a test power of 0.80) and statistical parametric mapping (SPM1D) to evaluate differences between control conditions. Subjects' kinetics, kinematics, muscle forces, and bone displacements were processed and analyzed using SPSS for Windows (version 25.0, SPSS Science Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects had experienced at least one acute sprain of the ankle joint.
* Those who experienced symptoms of pain and instability during daily activities or sports.
* No other serious diseases affecting the function of the lower limbs (e.g., arthritis, severe knee lesions, etc.).
* AOFAS < 80 points and VAS ≤ 3 on the affected side.
* The onset of injury is usually limited to 7 days to ensure that it is in the acute phase.
* Participants maintained a steady level of daily activity during the study period.

Exclusion Criteria:

* History of severe structural injury or surgery to the ankle (e.g., ligament reconstruction surgery, arthroscopic surgery, etc.).
* Presence of neuromuscular disease, or women during pregnancy.
* Allergy to muscle patch materials or history of skin disease. Ankle-related surgery or rehabilitation within the last 6 months.
* Before the initiation of data collection, all participants provided their written informed consent.

Ages: 18 Weeks to 44 Weeks | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Joint stiffness | four weeks
  Joint stiffness Δτ （change in torque）and Δθ （change in angle）will be combined to report Joint stiffness in Nm/rad

SECONDARY OUTCOMES:
Joint power | two weeks
  Τ(Joint moment) andω(Joint angular velocity) will be combined to report Joint Power in W/kg

CONTACTS AND LOCATIONS:
Overall Officials: dong yao gu, Principal Investigator — Ningbo University
Locations (1):
- Ningbo University, Zhejiang Province, Ningbo, China

IPD SHARING:
Plan to Share IPD: No
Data that contains information that can directly or indirectly identify an individual (such as rare diseases, geographic location, genetic data) must be strictly anonymized, otherwise it may violate the General Data Protection Regulation (GDPR) or the Health Insurance Portability and Accountability Act (HIPAA).

REFERENCES:
- [Derived] Wei Y, Xu D, Zhou Z, Qu X, Baker JS, Xiang L, Gu Y. The effects of kinesiology taping on joint stability during descending stairs in patients with acute ankle injuries. BMC Sports Sci Med Rehabil. 2025 Sep 25;17(1):271. doi: 10.1186/s13102-025-01321-0. PMID 40999475
- See also: Sarvestan, J, Svoboda Z, Linduška P, Hrasky P, Rutkowska-Kucharska A. The effect of ankle Kinesio™ taping on ankle joint biomechanics during unilateral balance status among collegiate athletes with chronic ankle sprain. Phys Ther Sport. 2020.45:161-167. — https://doi.org/10.1016/j.ptsp.2020.06.007